CLINICAL TRIAL: NCT02320435
Title: A Single-Arm Open-Label Multi-Centre Extension Study of Pertuzumab Administered As a Single Agent or in Combination With Other Anti-Cancer Therapies in Patients Previously Enrolled in a Hoffmann-La Roche-Sponsored Pertuzumab Study
Brief Title: A Safety and Efficacy Extension Study of Pertuzumab in Patients With Solid Tumors Previously Enrolled in a Hoffmann-La Roche-Sponsored Pertuzumab Clinical Trial
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO29406; 2014-002048-42 (EudraCT Number); 2023-505102-42-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pertuzumab (Single-Agent or Combination Therapy) (Experimental): Pertuzumab will continue to be administered as a single agent or in combination with other anti-cancer therapies at the same dose, schedule, and guidelines that were in effect at the end of the Parent study.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Other Combination Anti-Cancer Therapies

INTERVENTIONS:
Drug: Pertuzumab — In general, patients will continue to receive 420 milligrams (mg) of pertuzumab administered as an intravenous infusion every 3 weeks following the guidance of the Parent protocol.
  Other Names: RO4368451; Perjeta
Drug: Trastuzumab — If trastuzumab intravenous infusions were given in combination with pertuzumab as part of the Parent study, patients will continue to receive treatment at the same dose, schedule and under the same administration guidelines which were in effect at the time of Parent study closure.
Drug: Other Combination Anti-Cancer Therapies — If other anti-cancer therapies were given in combination with pertuzumab as part of the Parent study, patients will receive all treatments at the same dose, schedule and under the same administration guidelines which were in effect at the time of Parent study closure.

SUMMARY:
This is a single-arm, multi-center, open-label extension study designed to provide continued pertuzumab therapy to patients receiving pertuzumab as an investigational medicinal product (IMP) in a Roche-sponsored global study and who continue to receive pertuzumab at the end of the Parent study, as well as to collect long-term safety and efficacy data of pertuzumab therapy. Patients with solid tumors who have not experienced progressive disease in the Parent study and, in the investigator's opinion, may potentially benefit from continued pertuzumab treatment, will continue to receive pertuzumab until disease progression, unacceptable toxicity, investigator/patient decision, patient non-compliance, patient death, patient request to withdraw, or study termination by the Sponsor, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Prior eligibility for, and receiving pertuzumab as an investigational medicinal product in, a Roche-sponsored study (either as a single agent or in combination with other anti-cancer drugs used in the Parent study) at the time of the Parent study closure
* Investigator's opinion that the patient continues to benefit from treatment

Exclusion Criteria:

* Meets any of the exclusion criteria of the Parent protocol at the time the patient is considered for entry in the extension study
* Evidence of disease progression assessed according to Parent protocol before enrollment in to the extension study
* Permanent discontinuation of pertuzumab for any reason during the Parent study, or between the end of the Parent study and before enrollment into the extension study
* Any unresolved or irreversible toxicities during the Parent study that require permanent discontinuation of pertuzumab, according to Parent protocol or local label. Delay of treatment to wait for resolution of toxicities is allowed as long as it is within the guidelines of the respective Parent protocol and does not contradict exclusion criterion below.
* More than 9 weeks between the last dose of pertuzumab in the Parent study and the first dose pertuzumab in the extension study
* Left ventricular ejection fraction </= 50%
* Any serious uncontrolled concomitant disease that would contraindicate the use of pertuzumab or that would put the patient at high risk for treatment-related complications
* Treatment with any anti-cancer treatment (other than any treatment given as permitted in the Parent protocol) in the time period between last treatment in the Parent study and the first dose pertuzumab in the extension study (i.e. up to 9 weeks)
* Positive serum pregnancy test
* Women of child-bearing potential and men with partners of childbearing potential who do not agree to use a highly-effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the patient and/or partner for the duration of study treatment and for at least 7 months after the last dose of study medication. Male patients who do not agree to refrain from donating sperm during this same period. Male patients whose partner is pregnant who do not agree to use condoms for the duration of the pregnancy.
* Concurrent participation in any therapeutic clinical trial (other than the Parent study)
* Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of first dose of pertuzumab in this study until the date of disease progression or death, whichever occurs first (up to approximately 10 years)
Overall Survival | From date of first dose of pertuzumab in this study until the date of death (up to approximately 10 years)
Number of Participants with Adverse Events by Severity, Classified According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03 | From Baseline until 7 months after the last dose of pertuzumab (up to approximately 10 years)
Number of Participants with Adverse Events Leading to Pertuzumab Discontinuation or Dose Interruption | From Baseline until 7 months after the last dose of pertuzumab (up to approximately 10 years)
Number of Participants with Non-Serious Adverse Events of Special Interest (AESIs) | From Baseline until 7 months after the last dose of pertuzumab (up to approximately 10 years)
  Non-serious AESIs for this study include the following: Cases of potential drug-induced liver injury that include an elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's law; Suspected transmission of an infectious agent by the study drug; or, An asymptomatic decline in left ventricular ejection fraction (LVEF) requiring treatment or leading to discontinuation of human epidermal growth factor receptor 2 (HER2)-targeted therapies.
Left Ventricular Ejection Fraction (LVEF) Over Time | Baseline, every 3 treatment cycles (1 cycle is 21 days), and 28 days after last dose of pertuzumab (up to approximately 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (59):
- Brazil (8):
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo, São Paulo
  - Instituto de Oncologia de Sorocaba - CEPOS, Sorocaba, São Paulo
  - Instituto Nacional de Cancer - INCa, Rio de Janeiro
- China (8):
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning cancer Hospital & Institute, Shenyang
- Hospital Metropolitano (Sede Lindora-Santa Ana), San José, Costa Rica
- France (4):
  - Centre Georges Francois Leclerc, Dijon
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
- Germany (5):
  - Hämatologisch-Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus, Frankfurt am Main
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Praxis für Ambulante Onkologie im Krankenhaus Jerusalem, Hamburg
  - Studienzentrum UnterEms;Onkologische Schwerpunktpraxis Leer, Leer
  - Onkologische Praxis Neumarkt (Dr. med. Ekkehart Ladda), Neumarkt
- Italy (7):
  - Irccs Ist. Tumori Giovanni Paolo Ii, Bari, Apulia
  - Az. Osp. S. Orsola Malpighi, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - AUSL ? IRCCS Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - Asst Di Monza, Monza, Lombardy
  - A.O. Universitaria Pisana, Pisa, Tuscany
- Japan (3):
  - National Cancer Center Hospital East, Chiba
  - Gifu University Hospital, Gifu
  - Saitama Cancer Center, Saitama
- Mexico (3):
  - Iem-Fucam, D.F., Mexico CITY (federal District)
  - Cancerologia de Queretaro, Querétaro City, Querétaro
  - Instituto Nacional de Cancerologia, Distrito Federal
- Peru (3):
  - Hospital Nacional Carlos Alberto Seguin Escobedo-Essalud, Arequipa
  - Clinica Anglo Americana - Centro de Investigacion Oncologia CAA, Lima
  - Clinica Internacional, Sede San Borja, Lima
- Samodzielny Publiczny Kliniczny Nr 1 W Lublinie, Lublin, Poland
- Portugal (4):
  - IPO de Coimbra, Coimbra
  - Hospital da Luz, Lisbon
  - Hospital de Santa Maria, Lisbon
  - IPO do Porto, Porto
- Russia (2):
  - Kursk Regional Clinical Oncology Dispensary, Kursk
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- Ukraine (2):
  - Mun. Multifield Clin.Hosp.#4,Dept. of Chemotherapy, DSMU, Dnipropetrovsk
  - State Oncology Regional Treatment-Diagnostic Center, Lviv

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing